CLINICAL TRIAL: NCT03758144
Title: Rifaximin Improves Insulin Resistance in Metabolic Syndrome and Reduces Insulin Requirement in Type 2 Diabetes
Brief Title: Rifaximin Improves Gut Dysbiosis in Insulin Resistance and Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Amr Shaaban Hanafy, Assistant professor of medicine, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4493
Record Dates: First submitted 2018-11-16; First posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Type2 Diabetes
Keywords: gut dysbiosis; rifaximin; insulin resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study (Active Comparator)
  Interventions: Drug: Rifaximin 200 MG
- CONTROL GROUP (No Intervention)

INTERVENTIONS:
Drug: Rifaximin 200 MG — patients with type 2 diabetes and gut dysbiosis will be given rifaximin
  Arms: study

SUMMARY:
Gut Dysbiosis had been involved in some way in the pathogenesis of some extra-intestinal disorders including metabolic syndrome, cardiovascular disease, and obesity.

DETAILED DESCRIPTION:
Accumulating evidence had linked metabolic syndrome and diabetes to dysequilibrium in gut microbiota, which are a critical regulator of host metabolism and immune responses. gut microbiota interacts with host signaling pathways, leading to modulation of the endocrine system, immune responses. gut microbial metabolites, in particular, short-chain fatty acids, have been significantly associated with liability to diabetes. patients with positive fecal short-chain fatty acids will be given rifaximin

ELIGIBILITY:
Inclusion Criteria:

* diabetes with gut dysbiosis

Exclusion Criteria:

* recent antibiotic use
* pregnancy
* diabetogenic drugs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
change in glycemic control | 3 months
  Fasting blood sugar, post-prandial blood sugar (mg/dl)

SECONDARY OUTCOMES:
Gastrointestinal symptom questionnaire | 1 month
  symptomatic improvement in Dyspepsia, distension, abdominal pain

OTHER OUTCOMES:
change in weight | 6 months
  Weight loss in kilograms

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No
personal contact